CLINICAL TRIAL: NCT03558152
Title: A Phase II, Randomized, Parallel-Group, Double-Blind, Double-Dummy, Placebo-Controlled, Multicenter Study To Evaluate the Efficacy, Safety, and Pharmacokinetics of UTTR1147A Compared With Placebo and Compared With Vedolizumab in Patients With Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of UTTR1147A Compared With Placebo and With Vedolizumab in Participants With Moderate to Severe Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GA39925; 2017-002350-36 (EudraCT Number)
Record Dates: First submitted 2018-06-01; First posted 2018-06-15 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) (Experimental): Part A: UTTR1147A dose level 1 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: Vedolizumab Placebo
- Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) (Experimental): Part A: UTTR1147A dose level 1 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: UTTR1147A Placebo; Drug: Vedolizumab Placebo
- Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) (Experimental): Part A: UTTR1147A dose level 2 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: Vedolizumab Placebo
- Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) (Experimental): Part A: UTTR1147A dose level 2 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: UTTR1147A Placebo; Drug: Vedolizumab Placebo
- Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) (Experimental): Part A: UTTR1147A dose level 3 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: Vedolizumab Placebo
- Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) (Experimental): Part A: UTTR1147A dose level 3 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A; Drug: UTTR1147A Placebo; Drug: Vedolizumab Placebo
- Arm 4: Vedolizumab (Active Comparator): Parts A and B: Vedolizumab and UTTR1147A Placebo.
  Interventions: Drug: UTTR1147A Placebo; Drug: Vedolizumab
- Arm 5: Placebo (Placebo Comparator): Parts A and B: UTTR1147A Placebo and Vedolizumab Placebo.
  Interventions: Drug: UTTR1147A Placebo; Drug: Vedolizumab Placebo

INTERVENTIONS:
Drug: UTTR1147A — UTTR1147A will be administered intravenously (IV) at dose levels 1, 2, or 3 in Part A, and at the maintenance dose level in Part B, per the respective arm descriptions.
  Other Names: Efmarodocokin alfa; RO7021610; RG7880; IL-22Fc
  Arms: Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B); Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B); Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B); Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B); Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B); Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B)
Drug: UTTR1147A Placebo — The matching placebo to UTTR1147A (UTTR1147A Placebo) will be administered IV.
  Arms: Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B); Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B); Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B); Arm 4: Vedolizumab; Arm 5: Placebo
Drug: Vedolizumab — Vedolizumab will be administered IV, as specified in the prescribing information.
  Other Names: Entyvio
  Arms: Arm 4: Vedolizumab
Drug: Vedolizumab Placebo — The matching placebo to vedolizumab (Vedolizumab Placebo) will be administered IV.
  Arms: Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B); Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B); Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B); Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B); Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B); Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B); Arm 5: Placebo

SUMMARY:
This study is designed to evaluate the efficacy, safety, and pharmacokinetics of UTTR1147A compared with vedolizumab and with placebo in the treatment of participants with moderate to severe UC. This study will consist of two parts, Part A and Part B. Part A will test the induction of clinical remission and Part B will test the durability of clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of UC
* Confirmation of moderately to severely active UC, defined by the Mayo Clinic Score
* Inadequate response, loss of response, or intolerance to prior immunosuppressant treatment (i.e., azathioprine, 6-mercaptopurine, methotrexate, or tumor necrosis factor [TNF] inhibitors [maximum of 2 prior TNF inhibitors]) and/or corticosteroid treatment
* Use of highly effective contraception as defined by the protocol

Exclusion Criteria:

* History of psoriasis or psoriatic arthritis; any other inflammatory skin disorders requiring oral corticosteroids, immunosuppressants, or biological therapy within the previous year; or primary sclerosing cholangitis
* History of cancer as defined by the protocol
* Significant uncontrolled comorbidity, such as cardiac, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders (excluding UC)
* Prior extensive colonic resection, subtotal or total colectomy, or proctocolectomy, or planned surgery for UC
* Diagnosis of indeterminate colitis or granulomatous (Crohn's) colitis or toxic megacolon within 12 months prior to screening
* Suspicion of ischemic colitis, radiation colitis, or microscopic colitis
* Current fistula or history of fistula, pericolonic abscess and stricture (stenosis) of the colon
* History or current evidence of unresectable colonic mucosal dysplasia or history of high-grade colonic mucosal dysplasia
* Prior treatment with UTTR1147A
* Prior treatment with vedolizumab, etrolizumab, natalizumab, efalizumab, or any other anti-integrin agents
* Prior treatment with rituximab
* Use of prohibited therapies, as defined by the protocol, prior to randomization
* Congenital or acquired immune deficiency
* Evidence or treatment of infections or history of infections, as defined by the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (72):
- United States (2):
  - Carolina Digestive Diseases, Greenville, North Carolina
  - University of Utah School of Medicine; Gastroenterology Division, Salt Lake City, Utah
- Bulgaria (2):
  - MHAT Saint Karidad EAD, Plovdiv
  - Multiprofile Hospital for Active Treatment Hadji Dimitar OOD, Sliven
- LLC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Germany (5):
  - Gastroenterologische Spezialpraxis-Berlin-Karlshorst, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - St. Marien Krankenhaus; Med. Klinik, Ludwigshafen
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Ulm; Klinik für Innere Medizin II, Ulm
- Greece (2):
  - Iatriko Palaiou Falirou; Gastrointestinal Department, Palaió Fáliro
  - EUROMEDICA General Clinic of Thessaloniki; Gastroenterology Department, Thessaloniki
- Magyar Honvédség Egészségügyi Központ; Országos Haemophilia Központ, Budapest, Hungary
- Portiuncula Hospital, Ballinasloe, Co Galway, Ireland
- Shaare Zedek Medical Center; Bait Vagan, Jerusalem, Israel
- Italy (5):
  - Policlinico Universitario Campus Biomedico Di Roma, Rome, Lazio
  - Complesso Integrato Columbus, Rome, Lazio
  - ASST di Monza - Azienda Ospedaliera San Gerardo; U.O. Farmacia -Settore A - Corpo Posteriore, Monza, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - Azienda Ospedaliera Di Padova, Padua, Veneto
- ICS ARENSIA Exploratory Medicine, Chisinau, Moldova
- Poland (18):
  - SPZOZ Uniwersytecki SK nr 1 im N. Barlickiego UM w Lodzi; Oddz. Klin. Gastroenter. Og. i Onk., ?ód?
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy; Centrum Endoskopii Zabiegowej, Bydgoszcz
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Cz?stochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gda?sk
  - Synexus - Katowice, Katowice
  - Economicus - NZOZ ALL-MEDICUS; Zaklad Gastroenterologii, Katowice
  - ETG Kielce, Kielce
  - Gastromed SPK Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Klimed Marek Klimkiewicz, Piotrkow Trybunalski
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Późna
  - Clinical Research Center Sp. z o.o. MEDIC-R Spó?ka Komandytowa, Późna
  - Endoskopia Sp. z o.o., Sopot
  - Gastromed Kopon Zmudzinski i, Toru?
  - Centrum Zdrowia MDM, Warsaw
  - Jaroslaw Kierkus Prywatna Prakyka Lekarska, Warsaw
  - Przychodnia EuroMediCare, Wroc?aw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroc?aw
  - Melita Medical, Wroc?aw
- Russia (5):
  - Saint Martyr Elizabeth City Hospital, Saint Petersburg, Sankt-Peterburg
  - Irkutsk Research Centre Hospital of Siberian department of Russian Academy of Science, Irkutsk
  - Rostov State Medical University; Cardiorheumatology Department, Rostov-on-Don
  - North-West State Medical University n.a. I.I. Mechnikov, Saint Petersburg
  - Medical University Reaviz, Samara
- Serbia (7):
  - Clinical Hospital Center Zvezdara, Belgrade
  - KBC Dr Dragisa Misovic Dedinje, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Clinical Center Kragujevac; Clinic Of Psychiatry, Kragujevac
  - General Hospital Vrsac, Vršac
  - Clinical Hospital Centre Zemun, Zemun
  - General Hospital Djordje Joanovic - Zrenjanin, Zrenjanin
- Spain (2):
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Aparato Digestivo, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
- Ukraine (18):
  - Regional Municipal Institution Chernivtsi Regional Clinical Hospital; Gastroenterology department, Chernivtsi, Chernihiv Governorate
  - Medical Centre of PE First Private Clinic, Zhytomyr, Crimean Regional Governmenta
  - Ternopil University Hospital; Regional Center of Gastroenterology with Hepatology, Ternopil, Katerynoslav Governorate
  - City Clinical Hospital #1; Department of Gastroenterology, Vinnytsia, Kharkiv Governorate
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia, Kharkiv Governorate
  - ME Dnipropetrovsk Regional Clinical Hospital n.a. I.I Mechnykov Dnipropetrovsk Regional Council, Dnipro, KIEV Governorate
  - Treatment and Diagnostic Center of LLC MRT Elit, Kropyvnytskyi, KIEV Governorate
  - Medical Center of LLC Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Medical Center of Limited Liability Company ?Harmoniya krasy?, Kyiv, KIEV Governorate
  - Medical Center of LLC Medical Center Dopomoga Plus, Kyiv, KIEV Governorate
  - Medical Center of Edelweiss Medics LLC, Kyiv, KIEV Governorate
  - Synexus Affiliate - MC of LLC Medbud-Clinic, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - Medical Center of LLC Diaservis, Zaporizhzhia, KIEV Governorate
  - Clinic of SRI of Invalid Rehab. (ESTC) of VNMU n.a. M.I.Pyrohov, Vinnytsia, Podolia Governorate
  - Medical Center of LLC Medical Center Family Medicine Clinic; Endoscopy & Gastroenterology, Dnipr, Polissya Okruha
  - Transcarpathian Regional Clinical Hospital n.a. A. Novak; Rheumatology Department, Uzhhorod
  - Medical Center of Diaservice LLC; Division of clinical trials conduct, Department #3, Zaporizhzhia
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Danese S, Rothenberg ME, Lim JJ, Ding HT, McBride JM, Chen Y, Dash A, Mar JS, Keir M, Peyrin-Biroulet L, Panes J, Colombel JF, Feagan B, Valentine JF, Schreiber S. A Randomized Phase II Study of Efmarodocokin Alfa, an interleukin-22 Agonist, Versus Vedolizumab in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2025 Jul;23(8):1387-1397. doi: 10.1016/j.cgh.2024.11.013. Epub 2024 Dec 16. PMID 39694207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were assigned in a 1:1:1:1:1:1:2:1 ratio to one of eight treatment arms. Following completion of the screening period and after all patient eligibility requirements were confirmed, patients were assigned a patient number and randomly assigned to a treatment arm through an interactive voice or Web-based response system (IxRS).
Groups:
- Arm: 2A: UTTR1147A 60 + UTTR1147A; Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B): Part A: UTTR1147A dose level 3 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
- Arm: 2B: UTTR1147A 60 + Placebo: Part A: UTTR1147A dose level 2 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
- Arm 4: Vedolizumab: Participants received Vedolizumab and UTTR1147A Placebo
- Arm 5: Placebo: Participants received UTTR1147A Placebo and Vedolizumab Placebo.
Period: Overall Study
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm: 2A: UTTR1147A 60 + UTTR1147A | Arm: 2B: UTTR1147A 60 + Placebo | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Started | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Completed | 7 | 6 | 8 | 8 | 3 | 7 | 21 | 6
Not Completed | 15 | 15 | 13 | 15 | 19 | 14 | 22 | 16
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Rolled over in GA40209 due to worsening of disease | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscalculation in mmcs | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Mistake in calculation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Mistake in evaluation of disease status | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 1 | 1 | 1 | 3 | 2
Not completed — Lack of Efficacy | 11 | 11 | 10 | 11 | 14 | 12 | 14 | 13
Not completed — Protocol Violation | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Participants received UTTR1147A at a dose of 30 ug/kg
- Arm 2: Participants received UTTR1147A at a dose of 60 ug/kg
- Arm 3: Participants received UTTR1147A at a dose of 90 ug/kg
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo | Total
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (13.2) | 39.4 (12.1) | 39.5 (12.3) | 43.4 (14.8) | 41.9 (14.0) | 40.8 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 11 | 13 | 6 | 60
  Male | 28 | 29 | 32 | 30 | 16 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 43 | 44 | 43 | 43 | 22 | 195
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 43 | 43 | 43 | 43 | 22 | 194
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Remission at Week 8
Description: Clinical remission is defined as modified Mayo Clinic Score (mMCS) <= 2 with Mayo rectal bleeding subscore = 0, Mayo stool frequency subscore <=1 and Centrally read endoscopic score <= 1. Patients were classified as Non-Remitters if Week 8 assessments were missing or patient received permitted/ prohibited Rescue Therapy prior to assessment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Participants
  Yes | 5 | 4 | 5 | 11 | 2
  No | 38 | 40 | 38 | 32 | 20

2. Secondary Outcome: Percentage of Participants With Sustained Remission
Description: Sustained remission is defined as clinical remission at both Week 8 and Week 30, where clinical remission is defined as modified Mayo Clinic Score (mMCS) <= 2 with Mayo rectal bleeding subscore = 0, Mayo stool frequency subscore <=1 and Centrally read endoscopic score <= 1.
  Patients were classified as Non-Remitters at Week 8 or at Week 30 if assessments were missing or patient received permitted/prohibited Rescue Therapy prior to assessment
Time Frame: At Weeks 8 and 30
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Percentage of Participants | 4.55 [0.48 to 16.56] | 0.00 [0.00 to 10.38] | 0.00 [0.00 to 10.38] | 8.70 [2.34 to 21.52] | 4.55 [0.48 to 16.56] | 4.76 [0.50 to 17.29] | 20.93 [13.04 to 31.02] | 9.09 [2.44 to 22.42]

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of UTTR1147A
Time Frame: Days 1 - 29, Visit: Day 57
Population: Due to low enrollment in Part B of the study, the PK data from pooled Arms 1-3
  (1A + 1B; 2A + 2B; 3A + 3B) are summarized based on data up through Week 8 which is the primary efficacy assessment for Part A (Induction phase). A total of 130 patients who received at least one dose of efmarodocokin alfa and had measurable PK concentrations are included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 43 | 44 | 43
ng/mL
  Visit: Days 1 - 29 | 449 (658) | 590 (265) | 837 (560)
  Visit: Day 57: number analyzed (Participants) | 16 | 20 | 14
  Visit: Day 57 | 426 (344) | 693 (348) | 1340 (883)

4. Secondary Outcome: Minimum Serum Concentration (Cmin) of UTTR1147A
Time Frame: Days 1 - 29, Visit: Day 57
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 39 | 40 | 42
ng/mL
  Days 1 - 29 | 12.6 (9.55) | 28.3 (17.1) | 40.6 (27.7)
  Visit: Day 57: number analyzed (Participants) | 32 | 39 | 34
  Visit: Day 57 | 15.8 (11.7) | 37.2 (35.2) | 44.5 (28.1)

5. Secondary Outcome: Percentage of Participants With Clinical Response at Week 8
Description: Clinical response is defined as achieving clinical remission or as meeting both of the following criteria: A >= 3-point decrease from baseline in modified Mayo Clinic Score (mMCS); A >= 1-point decrease from baseline in rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.
  Patients were classified as Non-Responders if assessments were missing or patient received permitted/prohibited Rescue Therapy prior to assessment.
  NOTE: An Outcome Measure Description has not been entered.
Time Frame: At Week 8
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Percentage of Participants | 30.23 [20.99 to 40.95] | 36.36 [26.60 to 47.12] | 20.93 [13.04 to 31.02] | 53.49 [42.64 to 64.08] | 36.36 [22.48 to 52.27]

6. Secondary Outcome: Percentage of Participants With Clinical Response at Week 30
Description: Clinical response is defined as achieving clinical remission or as meeting both of the following criteria: A >= 3-point decrease from baseline in modified Mayo Clinic Score (mMCS); A >= 1-point decrease from baseline in rectal bleeding subscore or a rectal bleeding subscore of 0 or 1.
  Patients were classified as Non-Responders if assessments were missing or patient received permitted/prohibited Rescue Therapy prior to assessment.
Time Frame: At Week 30
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Percentage of Participants | 9.09 [2.44 to 22.42] | 4.76 [0.50 to 17.29] | 4.76 [0.50 to 17.29] | 13.04 [4.89 to 26.78] | 0.00 [0.00 to 9.94] | 4.76 [0.50 to 17.29] | 13.95 [7.50 to 23.21] | 0.00 [0.00 to 9.94]

7. Secondary Outcome: Percentage of Participants With Endoscopic Healing at Week 8
Description: Endoscopic healing is defined as a Mayo endoscopic subscore <= 1. Patients were classified as Non-Responders if assessments were missing or patient received permitted/prohibited Rescue Therapy prior to assessment.
Time Frame: At Week 8
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Percentage of Participants | 13.95 [7.50 to 23.21] | 13.64 [7.32 to 22.71] | 11.63 [5.77 to 20.51] | 32.56 [23.05 to 43.36] | 13.64 [5.12 to 27.89]

8. Secondary Outcome: Percentage of Participants With Endoscopic Healing at Week 30
Description: as for outcome 7
Time Frame: At Week 30
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Percentage of Participants | 13.64 [5.12 to 27.89] | 9.52 [2.56 to 23.40] | 14.29 [5.37 to 29.10] | 13.04 [4.89 to 26.78] | 4.55 [0.48 to 16.56] | 19.05 [8.58 to 34.52] | 30.23 [20.99 to 40.95] | 9.09 [2.44 to 22.42]

9. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 8
Description: Endoscopic remission is defined as a Mayo endoscopic subscore of 0. Patients were classified as Non-Responders if assessments were missing or patient received permitted/prohibited Rescue Therapy prior to assessment.
Time Frame: At Week 8
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Percentage of Participants | 4.65 [1.24 to 11.91] | 0.00 [0.00 to 5.10] | 4.65 [1.24 to 11.91] | 11.63 [5.77 to 20.51] | 0.00 [0.00 to 9.94]

10. Secondary Outcome: Percentage of Participants With Endoscopic Remission at Week 30
Description: as for outcome 9
Time Frame: At Week 30
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Percentage of Participants | 9.09 [2.44 to 22.42] | 4.76 [0.50 to 17.29] | 4.76 [0.50 to 17.29] | 13.04 [4.89 to 26.78] | 0.00 [0.00 to 9.94] | 4.76 [0.50 to 17.29] | 13.95 [7.50 to 23.21] | 0.00 [0.00 to 9.94]

11. Secondary Outcome: Change From Baseline in UC Bowel Movement Signs and Symptoms at Week 8, as Assessed by Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Score
Description: The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS). The bowel domain score ranges from 0-27, with a higher score indicating a worse disease state.
Time Frame: At Week 8
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Points on scale | -4.14 (5.06) | -6.39 (4.68) | -3.56 (6.11) | -6.23 (5.35) | -4.95 (5.70)

12. Secondary Outcome: Change From Baseline in UC Bowel Movement Signs and Symptoms at Week 30, as Assessed by Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Score
Description: as for outcome 11
Time Frame: At Week 30
Population: Number of analyzed participants reflects number of participants who submitted the EC-PRO questionnaire at Week 30.
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 5 | 6 | 7 | 7 | 1 | 5 | 20 | 5
Points on scale | -5.66 (7.92) | -3.62 (4.11) | -9.63 (5.15) | -6.63 (3.60) | -12.0 (NA) — No SD calculated as only 1 participant was analyzed. | -5.44 (9.47) | -8.32 (3.69) | -6.86 (5.32)

13. Secondary Outcome: Change From Baseline in UC Abdominal Signs and Symptoms at Week 8, as Assessed by Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Score
Description: The UC-PRO is being reported in three domains; two domains are key endpoints and reported as UC-PRO Signs and Symptoms (UC-PRO/SS). The functional (abdominal symptoms) domain score ranges from 0-12, with a higher score indicating a worse disease state.
Time Frame: At Week 8
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Points on scale | -0.96 (1.81) | -1.83 (1.76) | -1.82 (2.44) | -1.69 (2.25) | -1.15 (2.06)

14. Secondary Outcome: Change From Baseline in UC Abdominal Signs and Symptoms at Week 30, as Assessed by Ulcerative Colitis Patient-Reported Outcome Signs and Symptoms (UC-PRO/SS) Score
Description: as for outcome 13
Time Frame: At Week 30
Population: Number of analyzed participants reflects number of participants who submitted the EC-PRO questionnaire at Week 30.
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 0 | 4 | 17 | 5
Points on scale | -1.76 (3.21) | -0.64 (0.89) | -1.98 (2.06) | -1.05 (0.53) |  | -4.05 (1.96) | -1.82 (1.90) | -1.50 (3.60)

15. Secondary Outcome: Change From Baseline in Patient-Reported Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 8
Description: The IBDQ score is a Total Score summed up from across all 32 questions on the questionnaire. The Total Score range is from 32 to 224 with higher scores representing a better quality of life.
Time Frame: At Week 8
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Points on scale | 31.85 (39.64) | 31.95 (30.66) | 25.16 (40.00) | 44.85 (30.75) | 27.05 (41.35)

16. Secondary Outcome: Change From Baseline in Patient-Reported Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 30
Description: as for outcome 15
Time Frame: At Week 30
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Arm 1a: UTTR1147A Dose Level 1 (Part A) + UTTR1147A (Part B) | Arm 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B) | Arm 2a: UTTR1147A Dose Level 2 (Part A) + UTTR1147A (Part B) | Arm 2b: UTTR1147A Dose Level 2 (Part A) + Placebo (Part B) | Arm 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) | Arm 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B) | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21 | 43 | 22
Points on scale | 45.13 (28.62) | 35.50 (27.45) | 41.00 (23.28) | 41.38 (32.00) | 72.33 (19.35) | 55.43 (56.89) | 61.95 (34.75) | 53.00 (45.84)

17. Secondary Outcome: Percentage of Participants With Adverse Events
Time Frame: Up to 30 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4: Vedolizumab | Arm 5: Placebo
Number analyzed (Participants) | 43 | 44 | 43 | 43 | 22
Participants
  Non-Serious Adverse Events | 12 | 11 | 15 | 6 | 4
  Serious Adverse Events | 1 | 1 | 5 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Presence of Anti-Drug Antibodies (ADA) at Baseline and After Drug Administration
Time Frame: Baseline up to 30
Population: Participants in placebo groups were not analyzed for post-baseline Anti-Drug Antibodies (ADA)
Measure: Count of Participants; unit: Participants
Groups:
- Arm 1a; Arm 1B: Participants received UTTR1147A at a dose of 30 ug/kg
- Arm 2a; Arm 2b: Participants received UTTR1147A at a dose of 60 ug/kg
- Arm 3a; Arm 3b: Participants received UTTR1147A at a dose of 90 ug/kg
Arm/Group | Arm 1a | Arm 1B | Arm 2a | Arm 2b | Arm 3a | Arm 3b
Number analyzed (Participants) | 22 | 21 | 21 | 23 | 22 | 21
Participants | 0 | 2 | 1 | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 30 weeks
Description: Only patients who meet the criteria for clinical response at Week 8 (the end of induction phase, without use of rescue therapy) continued into the maintenance phase.
Groups:
- Arm 1: UTTR1147A 30 ug/kg Induction: Combined arms: 1A: UTTR1147A 30 + UTTR1147A and 1b: UTTR1147A Dose Level 1 (Part A) + Placebo (Part B)
- Arm 2: UTTR1147A 60 ug/kg Induction: Combined arms: 2A: UTTR1147A 60 + UTTR1147A and 2B: UTTR1147A 60 + Placebo
- Arm 3: UTTR1147A 90 ug/kg Induction: Combined arms: 3a: UTTR1147A Dose Level 3 (Part A) + UTTR1147A (Part B) and 3b: UTTR1147A Dose Level 3 (Part A) + Placebo (Part B)
- Arm 4: VEDOLIZUMAB 300 mg Induction; ARM4: VEDOLIZUMAB 300 + VEDOLIZUMAB 300Maintenance: Parts A and B: Vedolizumab and UTTR1147A Placebo.
- Arm 5: PLACEBO Induction; ARM5: PLACEBO + PLACEBOMaintenance: Parts A and B: UTTR1147A Placebo and Vedolizumab Placebo.
- 1A: UTTR1147A 30 + UTTR1147A 60Maintenance: Part A: UTTR1147A dose level 1 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
- 1B: UTTR1147A 30 + PLACEBOMaintenance: Part A: UTTR1147A dose level 1 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
- 2A: UTTR1147A 60 + UTTR1147A 60Maintenance; 3A: UTTR1147A 90 + UTTR1147A 60Maintenance: Part A: UTTR1147A dose level 3 and Vedolizumab Placebo.
  Part B: UTTR1147A maintenance dose and Vedolizumab Placebo.
- 2B: UTTR1147A 60 + PLACEBOMaintenance: Part A: UTTR1147A dose level 2 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
- 3B: UTTR1147A 90 + PLACEBOMaintenance: Part A: UTTR1147A dose level 3 and Vedolizumab Placebo.
  Part B: UTTR1147A Placebo and Vedolizumab Placebo.
Arm/Group | Arm 1: UTTR1147A 30 ug/kg Induction | Arm 2: UTTR1147A 60 ug/kg Induction | Arm 3: UTTR1147A 90 ug/kg Induction | Arm 4: VEDOLIZUMAB 300 mg Induction | Arm 5: PLACEBO Induction | 1A: UTTR1147A 30 + UTTR1147A 60Maintenance | 1B: UTTR1147A 30 + PLACEBOMaintenance | 2A: UTTR1147A 60 + UTTR1147A 60Maintenance | 2B: UTTR1147A 60 + PLACEBOMaintenance | 3A: UTTR1147A 90 + UTTR1147A 60Maintenance | 3B: UTTR1147A 90 + PLACEBOMaintenance | ARM4: VEDOLIZUMAB 300 + VEDOLIZUMAB 300Maintenance | ARM5: PLACEBO + PLACEBOMaintenance
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 1/43 | 0/43 | 0/22 | 0/10 | 0/7 | 0/10 | 0/9 | 0/6 | 0/8 | 0/22 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/44 | 5/43 | 0/43 | 0/22 | 0/10 | 0/7 | 0/10 | 0/9 | 0/6 | 0/8 | 0/22 | 0/7
Other Adverse Events (participants affected / at risk) | 12/43 | 11/44 | 15/43 | 6/43 | 4/22 | 2/10 | 2/7 | 6/10 | 3/9 | 2/6 | 3/8 | 2/22 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: UTTR1147A 30 ug/kg Induction (N=43) | Arm 2: UTTR1147A 60 ug/kg Induction (N=44) | Arm 3: UTTR1147A 90 ug/kg Induction (N=43) | Arm 4: VEDOLIZUMAB 300 mg Induction (N=43) | Arm 5: PLACEBO Induction (N=22) | 1A: UTTR1147A 30 + UTTR1147A 60Maintenance (N=10) | 1B: UTTR1147A 30 + PLACEBOMaintenance (N=7) | 2A: UTTR1147A 60 + UTTR1147A 60Maintenance (N=10) | 2B: UTTR1147A 60 + PLACEBOMaintenance (N=9) | 3A: UTTR1147A 90 + UTTR1147A 60Maintenance (N=6) | 3B: UTTR1147A 90 + PLACEBOMaintenance (N=8) | ARM4: VEDOLIZUMAB 300 + VEDOLIZUMAB 300Maintenance (N=22) | ARM5: PLACEBO + PLACEBOMaintenance (N=7)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: UTTR1147A 30 ug/kg Induction (N=43) | Arm 2: UTTR1147A 60 ug/kg Induction (N=44) | Arm 3: UTTR1147A 90 ug/kg Induction (N=43) | Arm 4: VEDOLIZUMAB 300 mg Induction (N=43) | Arm 5: PLACEBO Induction (N=22) | 1A: UTTR1147A 30 + UTTR1147A 60Maintenance (N=10) | 1B: UTTR1147A 30 + PLACEBOMaintenance (N=7) | 2A: UTTR1147A 60 + UTTR1147A 60Maintenance (N=10) | 2B: UTTR1147A 60 + PLACEBOMaintenance (N=9) | 3A: UTTR1147A 90 + UTTR1147A 60Maintenance (N=6) | 3B: UTTR1147A 90 + PLACEBOMaintenance (N=8) | ARM4: VEDOLIZUMAB 300 + VEDOLIZUMAB 300Maintenance (N=22) | ARM5: PLACEBO + PLACEBOMaintenance (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 (6) | 1 (2) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Herpes zoster infection neurological (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (4) | 3 (6) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 1 (2) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (8) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 2 (6) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (6) | 5 (14) | 9 (28) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT03558152/Prot_SAP_000.pdf